CLINICAL TRIAL: NCT05329116
Title: Efficacy of Mesotherapy Added to Intra-articular Platelet-rich Plasma (PRP) in Patients
Brief Title: Efficacy of Mesotherapy Added to Intra-articular Platelet-rich Plasma (PRP) in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Necmettin Yildiz (Other)
Responsible Party: Sponsor-Investigator, Necmettin Yildiz, Clinical Professor, Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PamukkaleU-Simsek-001
Record Dates: First submitted 2022-03-23; First posted 2022-04-14 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Osteo Arthritis Knee
Keywords: Mesotherapy; Platelet-Rich Plasma; Osteo Arthritis Knee
MeSH Terms: interventions — Lidocaine; Pentoxifylline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-articular PRP (Active Comparator): For PRP treatment, 8 mL of peripheral blood will be taken from the patient and centrifuged at 4000 rpm for 8 minutes. Then, 3-4 mL of PRP will be taken and used for intra-articular injection. Patients will receive a single session of PRP treatment.
  Interventions: Biological: Platelet-rich plasma
- Intra-articular PRP + periarticular mesotherapy (Active Comparator): In addition to single session PRP treatment, patients will receive 3 weeks of mesotherapy treatment once a week (the first session will be with PRP treatment).
  Sterile and disposable needle tip (0.26mm × 4mm and 0.3mm × 13 mm, Terumo) will be used in mesotherapy. Patients will be administered 1.5 ml of 2% lidocaine, 1.5 ml of 30 mg of pentoxifylline.
  Among the injection techniques, profundal intradermic injection (IDP, injection depth: 2-4 mm) and superficial intradermic injection (IDS, injection depth: 1-2 mm) will be used.
  Interventions: Drug: Lidocaine 2% Injectable Solution; Biological: Platelet-rich plasma

INTERVENTIONS:
Drug: Lidocaine 2% Injectable Solution — Patients will be administered 1.5 ml of 2% lidocaine, 1.5 ml of 30 mg of pentoxifylline.
  Among the injection techniques, profundal intradermic injection (IDP, injection depth: 2-4 mm) and superficial intradermic injection (IDS, injection depth: 1-2 mm) will be used.
  8 mL of peripheral blood will be taken from the patient and centrifuged at 4000 rpm for 8 minutes. Then, 3-4 mL of PRP will be taken and used for intra-articular injection
  Other Names: pentoxifylline
  Arms: Intra-articular PRP + periarticular mesotherapy
Biological: Platelet-rich plasma — 8 mL of peripheral blood will be taken from the patient and centrifuged at 4000 rpm for 8 minutes. Then, 3-4 mL of PRP will be taken and used for intra-articular injection

SUMMARY:
In this study, the investigators aimed to determine whether platelet rich plasma (PRP) and mesotherapy combined treatment is effective on pain and function compared to PRP alone in patients with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
42 patients diagnosed with knee OA according to the criteria of the American College of Rheumatology (ACR) (15) who applied to Physical Medicine and Rehabilitation outpatient clinic will be recruited. Patients' age, gender, occupation, medications, duration of diagnosis, body mass index, comorbidity, functional status and pain will be questioned.

After the participants are informed about the study, their consent will be obtained.

Patients will be randomized using a random numbers table. The first group will receive intra-articular PRP therapy. The second group will receive mesotherapy treatment in addition to PRP treatment.

Group 1: Intra-articular PRP:

For PRP treatment, 8 mL of peripheral blood will be taken from the patient and centrifuged at 4000 rpm for 8 minutes. Then, 3-4 mL of PRP will be taken and used for intra-articular injection (16). Patients will receive a single session of PRP treatment.

Group 2: Intra-articular PRP + periarticular mesotherapy In addition to single session PRP treatment, patients will receive 3 weeks of mesotherapy treatment once a week (the first session will be with PRP treatment).

Sterile and disposable needle tip (0.26mm × 4mm and 0.3mm × 13 mm, Terumo) will be used in mesotherapy. Patients will be administered 1.5 ml of 2% lidocaine, 1.5 ml of 30 mg of pentoxifylline.

Among the injection techniques, profundal intradermic injection (IDP, injection depth: 2-4 mm) and superficial intradermic injection (IDS, injection depth: 1-2 mm) will be used (14).

All patients will be evaluated with the following evaluation parameters before the treatment, at the 1st month and at the 3rd month after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-80 years
* To be diagnosed with knee OA according to the diagnosis of ACR
* Ability to give informed consent

Exclusion Criteria:

* History or symptoms of lower extremity surgery, ligament injury, balance disorder or lower extremity injury in the last 6 months
* Allergic to lidocaine, other local anesthetics and pentoxifylline
* Intra and periarticular injection in the last 3 months
* Use of NSAIDs for pain relief in the past 7 days
* Presence of local or systemic infection
* cancer history
* Heart failure, cardiac arrhythmia
* Bleeding diathesis, antiaggregant, anticoagulant use
* Cerebral hemorrhage
* Pregnancy or breastfeeding
* Presence of psychiatric or neurological disease affecting cooperation, cognitive and neurological functions
* Inability to complete the survey

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-12-25 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from Baseline VAS at 1st month after the treatment.
  The pain score will be measured using a 10 cm millimetric visual analog scale (VAS), where patients are asked to mark the degree of pain intensity from 0 (no pain) to 10 (worst pain imaginable) before and after treatment.
Visual Analogue Scale (VAS) | Change from Baseline VAS at 3rd month after the treatment.
  The pain score will be measured using a 10 cm millimetric visual analog scale (VAS), where patients are asked to mark the degree of pain intensity from 0 (no pain) to 10 (worst pain imaginable) before and after treatment.
Visual Analogue Scale (VAS) | Change from 1st month VAS at 3rd month after the treatment.
  The pain score will be measured using a 10 cm millimetric visual analog scale (VAS), where patients are asked to mark the degree of pain intensity from 0 (no pain) to 10 (worst pain imaginable) before and after treatment.

SECONDARY OUTCOMES:
WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) | at the 1st and the 3rd months after the treatment.
  The evaluation of pain, stiffness and physical functions of the patients included in the study before and after treatment will be made using the Turkish version of the WOMAC criterion. WOMAC is a specific, valid and reliable criterion for OA and includes 24 questions under three sub-headings: pain, stiffness and physical function. Each question was scored on a Likert scale as 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe. The score of each section is calculated on its own and the total score ranges from 0 to 100. High scores indicate increased pain and stiffness and impaired physical function.
Range of Motion (ROM) | at the 1st and the 3rd months after the treatment.
  The normal ROM of the knee is 135 degrees in flexion and 0 in extension. The knee ROM of the patients included in the study will be measured and recorded before and after the treatment.
Side Effect | at the 1st and the 3rd months after the treatment.
  Side effects observed at the end of treatment in both groups will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No